CLINICAL TRIAL: NCT01880866
Title: An Open Label Pilot Study of Purified (-)-Epicatechin to Improve Hemodynamics in Pulmonary Arterial Hypertension
Brief Title: (-)-Epicatechin and Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI
Record Dates: First submitted 2013-05-28; First posted 2013-06-19 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Catechin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (-)-Epicatechin (Experimental): A single dose of 100mg or 200mg (-)-Epicatechin to be administered orally
  Interventions: Drug: (-)-Epicatechin

INTERVENTIONS:
Drug: (-)-Epicatechin — A single dose of purified (-)-epicatechin will be administered orally to subjects after a regularly scheduled right heart catheterization. The subjects will be monitored for 5 hours and released.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a progressive disease that results in severe activity limitation and death. There are few treatments for PAH and the available medications are expensive, difficult to administer and have significant toxicities.

(-)-Epicatechin is a non-toxic compound that naturally occurs in foods such as tea, wine and chocolate. Clinical intervention studies using dark chocolate in normal volunteers and subjects at risk for or with established cardiovascular disease have demonstrated improvements in peripheral and coronary vascular endothelial function, blood pressure, lipids, glucose tolerance and inflammatory markers.

Our study intends to examine the hemodynamics effects of purified (-)-epicatechin in subjects with pulmonary arterial hypertension. We hypothesize purified (-)-epicatechin will reduce pulmonary vascular resistance in patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 or older
* NYHA Class II-!V
* 6 minute walk distance < 450 meters
* Outpatients with suspected WHO group I PAH or and established diagnosis of WHO group I PAH undergoing clinically indicated right heart catheterization
* Written informed consent obtained from subject and ability for subject to comply with the requirements of study

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Systolic blood pressure <100 or >160
* History of migraine headaches
* Allergy or intolerance to chocolate, tea or wine
* Subject is considered unsuitable for the study in the opinion of the investigator, nurse practitioner, or study physician for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Resistance Index | up to 5 hours after right heart catheterization
  This study will assess acute hemodynamic effects, specifically effects on pulmonary vascular resistance index (PVRI), of a single dose of purified (-)-epicatechin in patients with patients with PAH.

SECONDARY OUTCOMES:
Endothelial function and hemodynamics | up to 5 hours after right heart catheterization
  Secondary objectives are to determine if endothelial function, right heart function, nitric oxide and mitochondrial function improve following consumption of purified (-)-epicatechin.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barnett, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States